CLINICAL TRIAL: NCT07233551
Title: Utilization of CBC-Derived Inflammatory Indices in Assessing Severity and Prognosis of Acute Pancreatitis.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelhameed Ahmed Abdelhameed, Resident physician of internal medicine in Assiut university hospitals, Assiut University
Other Study IDs: AP Prognosis with IF indices
Record Dates: First submitted 2025-09-16; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Acute Pancreatitis (AP); Inflammatory Indices
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CBC derived inflammatory indices — Complete blood count, CBC_based inflammatory indices:
  1. Prognostic nutritional index (PNI):
     PNI is a score based on serum albumin and lymphocyte count, used to assess nutritional and immune status.
  2. Systemic inflammation response index (SIRI) :
     SIRI is an inflammatory marker used to assess systemic inflammation and predict prognosis in various diseases, including cancer and acute conditions.
  3. Systemic immune inflammation index (SII) :
     SII is a composite marker reflecting the balance between host immune and inflammatory status. It is widely used as a prognostic indicator in cancers, cardiovascular disease, and acute inflammatory conditions.
  4. platelet lymphcyte ratio (PLR) : (PLR) reflects the balance between thrombosis/inflammation (platelets) and immune regulation (lymphocytes).
  5. Neutrophile to lymphcyte ratio (NLR) :
  (NLR) is a widely used inflammatory marker derived from CBC, indicating systemic inflammation and immune response.

SUMMARY:
Utilization of CBC-Derived Inflammatory Indices in Assessing Severity and Prognosis of Acute Pancreatitis.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is a common disease that develops swiftly and has a mortality rate between 1% and 1.5%.

Investigators should therefore identify the severity of AP and the presence of complications early in order to reduce the risk of premature death and devise interventions to reduce mortality. Currently, the majority of conventional methods for assessing the severity of acute pancreatitis have limitations; the majority of these methods are insufficiently basic, rapid, and cost-effective. None of these methods are sufficiently sensitive or specific.

When acute pancreatitis occurs, trypsin is released and the exocrine function of the pancreas is activated, which destroys the pancreatic self-defence mechanism and exacerbates the damage and destruction of pancreatic cells. Consequently, the vascular endothelium is compromised, motor dystonia develops, vascular permeability increases, more leukocytes migrate to tissues, and coagulation systems are activated. Numerous inflammatory markers based on blood cell changes that were inexpensive and easily obtained during the early stages of hospitalisation were used to determine the severity of AP, including the red cell distribution width (RDW), neutrophil-lymphocyte ratio (NLR), lymphocyte-monocyte ratio (LMR), platelet lymphocyte ratio (PLR), total calcium (TC), albumin-corrected calcium (ACC), and blood urea nitrogen (BUN). However, there is little literature that compares their predictive functions comprehensively.

Because inflammatory mediators play a crucial role in the occurrence of AP, numerous inflammatory markers have recently been used to predict the prognosis of AP. SII is one of the new inflammatory markers that indicates the immune status. SII is a measure of systemic immune-inflammation based on neutrophils, lymphocytes, and platelets. SII was previously only associated with the prognosis of cancer patients; however, it has recently been applied to inflammation-related diseases.

In patients with severe acute pancreatitis (AP), numerous pancreatic cells are damaged, and as a result, inadequate insulin secretion can result in stressful fluctuations in blood glucose level. Blood glucose fluctuations are believed to cause irreversible organ injury and impact patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients aged 18 years old or older.
2. patients with acute pancreatitis who were treated in our hospital from January 2019 to March 2025.

Exclusion Criteria:

1. history of chronic kidney disease
2. Pregnancy.
3. History of neoplasm
4. present of acute infection
5. history of hematological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with AP who were treated in our hospital (Al Rhaghe hospital) from January 2019 to March 2025 (age ≥18 years old; written consent will be obtained); also, we prospectively will analyse data of patients with AP who will be admitted within one year
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between Prognostic Nutritional Index (PNI) and Clinical Severity of Acute Pancreatitis | Between 48 and 72 hours after hospital admission
  PNI will be calculated as: PNI = 10 × serum albumin (g/dL) + 0.005 × total lymphocyte count (/mm³). The correlation between PNI (numeric value) and the clinical severity of acute pancreatitis (based on the Revised Atlanta Classification) will be assessed
Correlation between Systemic Immune-Inflammation Index (SII) and Clinical Severity of Acute Pancreatitis | Between 48 and 72 hours after hospital admission
  SII will be calculated as: SII = (Platelet count × Neutrophil count) / Lymphocyte count. The correlation between SII (numeric value) and clinical severity will be assessed.
Correlation between Systemic Inflammation Response Index (SIRI) and Clinical Severity of Acute Pancreatitis | Between 48 and 72 hours after hospital admission
  SIRI will be calculated as: SIRI = (Neutrophil count × Monocyte count) / Lymphocyte count. The correlation between SIRI (numeric value) and clinical severity will be assessed.
Correlation between Platelet-to-Lymphocyte Ratio (PLR) and Clinical Severity of Acute Pancreatitis | Between 48 and 72 hours after hospital admission
  PLR will be calculated as: PLR = Platelet count / Lymphocyte count. The correlation between PLR (numeric ratio) and clinical severity will be assessed.
Correlation between Neutrophil-to-Lymphocyte Ratio (NLR) and Clinical Severity of Acute Pancreatitis | Between 48 and 72 hours after hospital admission
  NLR will be calculated as: NLR = Neutrophil count / Lymphocyte count. The correlation between NLR (numeric ratio) and clinical severity will be assessed

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu W, Zhang Y, Zhang Y, Qu X, Zhang Z, Zhang R. Association Between the Systemic Inflammation Response Index and Severity of Acute Pancreatitis: A Retrospective Cohort Study. J Inflamm Res. 2025 Mar 27;18:4471-4480. doi: 10.2147/JIR.S512553. eCollection 2025. PMID 40166595
- [Background] Alzarea AI, Khan YH, Alanazi AS, Butt MH, Almalki ZS, AlAhmari AK, Alsahali S, Mallhi TH. Barriers and Facilitators of Pharmacoeconomic Studies: A Review of Evidence from the Middle Eastern Countries. Int J Environ Res Public Health. 2022 Jun 27;19(13):7862. doi: 10.3390/ijerph19137862. PMID 35805521
- [Background] Mirzaei-Alavijeh M, Amini M, Moradinazar M, Eivazi M, Jalilian F. Disparity in cognitive factors related to cancer screening uptake based on the theory of planned behavior. BMC Cancer. 2024 Jul 16;24(1):845. doi: 10.1186/s12885-024-12607-w. PMID 39014335
- [Background] Krinsley JS, Rule P, Pappy L, Ahmed A, Huley-Rodrigues C, Prevedello D, Preiser JC. The Interaction of Acute and Chronic Glycemia on the Relationship of Hyperglycemia, Hypoglycemia, and Glucose Variability to Mortality in the Critically Ill. Crit Care Med. 2020 Dec;48(12):1744-1751. doi: 10.1097/CCM.0000000000004599. PMID 33031146
- [Background] Lu Y, Zhang Q, Lou J. Blood glucose-related indicators are associated with in-hospital mortality in critically ill patients with acute pancreatitis. Sci Rep. 2021 Jul 28;11(1):15351. doi: 10.1038/s41598-021-94697-1. PMID 34321549
- [Background] Kim Y, Choi H, Jung SM, Song JJ, Park YB, Lee SW. Systemic immune-inflammation index could estimate the cross-sectional high activity and the poor outcomes in immunosuppressive drug-naive patients with antineutrophil cytoplasmic antibody-associated vasculitis. Nephrology (Carlton). 2019 Jul;24(7):711-717. doi: 10.1111/nep.13491. Epub 2019 Apr 29. PMID 30203901
- [Background] Liu G, Tao J, Zhu Z, Wang W. The early prognostic value of inflammatory markers in patients with acute pancreatitis. Clin Res Hepatol Gastroenterol. 2019 Jun;43(3):330-337. doi: 10.1016/j.clinre.2018.11.002. Epub 2018 Dec 10. PMID 30545732
- [Background] Gorgel SN, Akin Y, Koc EM, Kose O, Ozcan S, Yilmaz Y. Retrospective study of systemic immune-inflammation index in muscle invasive bladder cancer: initial results of single centre. Int Urol Nephrol. 2020 Mar;52(3):469-473. doi: 10.1007/s11255-019-02325-9. Epub 2019 Oct 28. PMID 31659597
- [Background] Peery AF, Crockett SD, Murphy CC, Lund JL, Dellon ES, Williams JL, Jensen ET, Shaheen NJ, Barritt AS, Lieber SR, Kochar B, Barnes EL, Fan YC, Pate V, Galanko J, Baron TH, Sandler RS. Burden and Cost of Gastrointestinal, Liver, and Pancreatic Diseases in the United States: Update 2018. Gastroenterology. 2019 Jan;156(1):254-272.e11. doi: 10.1053/j.gastro.2018.08.063. Epub 2018 Oct 10. PMID 30315778